CLINICAL TRIAL: NCT00204204
Title: The Multitraumatized Patient. What is the Importance of Forces Involved and the Use of Safety Equipment for the Amount of Trauma to the Patient Inside the Vehicle.
Brief Title: Importance of Forces and Safety Features in Car Crash Multitrauma
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Royal Department of Transportation (Unknown); Ullevaal University Hospital (Other); Health Region East, Norway (Other); Norwegian Air Ambulance Foundation (Other)
Other Study IDs: 216-05-04273; 200500715-2
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Multiple Trauma
Keywords: multiple trauma; traffic accident; outcome; safety; injury severity
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The pupose of the study is a prospective evaluation of external and internal factors/causes of importance for the trauma and final outcome experienced by persons inside motor vehicles in serious car accidents. We hypothesise that there is an association between the use and function of safety features and the results for the patient and an association between material damage and the severity of injury.

DETAILED DESCRIPTION:
We plan to study approximately 200 road accidents with multitraumatised patients and accidents with modern cars and severe material damage with little or moderate damage to persons inside the vehicle. A researcher will be alerted by the call centre (Norwegian 911-equivalent), move to the place of accident and take a pure observers role (unless ethically unacceptable due to lack of other health personnel). He will document the accident including use and condition of safety features, conditions inside the coupe, weather conditions, etc. Other available information on the vehicles, crashtests etc will be gathered from the manufacturer. All medical information will be gathered from the ambulance service, hospitals, pathology and forensic departments. Information from police and fire department will also be gathered.

Patient, next-of-kin, others invloved will be interviewed as appropriate in follow-up.

Four accident groups: Front-to-front or -object > 60 km/hour, same < 60 km/hour, car rolled over on road, car rolled over out-of-road. Factors: Age of vehicle, damage to coupe, cause of accident, on-scene time, initial evaluation by health personnel, injury severity scoring in hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple trauma from severe motor vehicle accidents in Eastern Norway patients from motor vehicle accidents in Eastern Norway with severe material damage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ulleval University Hospital, Oslo, Norway